CLINICAL TRIAL: NCT06087367
Title: Building of a Diagnostic/Prognostic Database by High-throughput Multiplexed Assays for Human ERG Variant Effects
Brief Title: Building of a Diagnostic/Prognostic Database for Human ERG Variant Effects
Acronym: CarDiag
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0456
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Long QT Syndrome
Keywords: Long QT syndrome; KCNH2 gene variants
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac channelopathies induce severe heart rhythm or conduction disorders. Mutations of the KCNH2 gene, that encodes the human (h) ERG channel, is responsible for 30-40% of all cases of long QT syndrome (inherited LQT2). Besides, hERG is frequently responsible for off-target effects of several pharmacological agents (acquired LQT2). With the advent of Next Generation Sequencing, hundreds of new KCNH2 variants are accumulating in regional databases including those developed by french centers of references. Worldwide, we estimate there are more than 1000 variants for hERG channel. Unfortunately, many of these new variants appear to be of unknown functional significance in spite of available clinical and genetic information. Little is known on whether they affect the channel biophysical properties, its expression at the cell surface and/or its structure. Yet, this information is crucial to determine the real degree of pathogenicity of these variants, and therefore to make the proper diagnosis on inherited LQT2, counsel the patient for his treatment and improve the management of the patient's life. Our ambition is therefore to tackle this issue of variant significance by (i) launching a large-scale multi-functional evaluation of hERG variants, (ii) introducing for the first time a formatted large-scale pathogenicity annotation score for all variants that have been functionally evaluated by this multi-parametric approach, and (iii) regrouping all the relevant information collected in every French Regional centers of reference into a single National database hosted by an infrastructure that possesses enough flexibility for continuous data implementation and cross-referencing. The database will integrate the latest International guidelines for functional pathogenicity annotation. This project will also include the pharmacological characterization of several drugs susceptible to produce acquired LQT2 with variable severities. We aim to understand whether there are structural regions within hERG channel in which the introduction of a variant is more prone to increase the risk of acquired LQT2 or if, on the contrary, a set of variants may relatively protect some patients against LQT2-inducing drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients carrier of a mutation in KCNH2 gene

Exclusion Criteria:

* Patients who refuse to take part to research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A collective effort will be conducted by all partners on identifying sets of priorities for KCNH2 variants. Priority 1 will be all the variants for which clinical and genetic data cannot decide on their own about the pathogenicity. All French variants will be included in this group. It may be enlarged by interesting variants identified from Clinvar. Priority 2 variants will be those for which pathogenicity is established but for which additional functional, pharmacological and structural data may be of interest. Special mention will be attributed to the variants that localize on hERG regions well defined structurally. Priority 3 are all other variants.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
To develop a database listing KCNH2 variants and their clinical impact | 42 months
  Biophysical and pharmacological characterization; Trafficking impact of hERG variants; Structural impact of hERG variants using modeling tools

SECONDARY OUTCOMES:
To stratify KCNH2 gene variants according to their sensitivity to drugs | 42 months
  Stratify KCNH2 gene variants according to their sensitivity to drugs known to induce acquired type 2 long QT syndrome

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nantes university hospital, Nantes, Loire-atlantique
  - Hôpital Bichat - Claude Bernard, Paris

IPD SHARING:
Plan to Share IPD: Yes
Implementation of a new web-accessible variant-centric database